CLINICAL TRIAL: NCT04962620
Title: Multicenter Prospective Non-interventional Study of the Efficacy and Safety of Longidaze®, Vaginal and Rectal Suppositories, 3000 IU, for the Treatment of Patients With External Genital Endometriosis
Brief Title: Study of the Efficacy and Safety of Longidaze® for the Treatment of Patients With External Genital Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Other Study IDs: ISLAND
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: External Genital Endometriosis
Keywords: longidaze; external genital endometriosis; bovhyaluronidase azoximer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Longidaze: 75 patients receiving combination therapy: Longidaze + dienogest
  Interventions: Drug: Bovhyaluronidase azoximer
- Control: 74 patients receiving only Dienogest.

INTERVENTIONS:
Drug: Bovhyaluronidase azoximer — Rectally or vaginally 1 suppository of Longidaze every 2 days. The main course of treatment - 10 suppositories (for 30 days). Then (according to the doctor's decision) supportive therapy is prescribed for 1 suppository 1 time in 7 days. Course of supportive treatment - 17 suppositories for another 120 days. The patients took dienogest according to the instructions for use.
  Groups: Longidaze

SUMMARY:
A study is being conducted to evaluate the efficacy and safety of Longidaze for the prevention and treatment of external genital endometriosis .

DETAILED DESCRIPTION:
The aim of the study is to compare the outcomes of complex therapy in patients with external genital endometriosis who, in addition to hormonal therapy, were prescribed Longidaze®, vaginal and rectal suppositories, 3000 IU, with the outcomes of therapy in patients who received only hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Documented informed consent;
2. Patients over 18 years of age with active menstrual function;
3. Women with external genital endometriosis, confirmed morphologically and visually during laparoscopic or laparotomy surgery performed 10 years to 2 weeks prior to Day 0;
4. Patients in the framework of routine clinical practice in accordance with the instructions for use, prior to inclusion in the study, are assigned one of the following therapy regimens:

   * monotherapy with dienogest 2 mg daily for at least 6 months per os
   * complex treatment with dienogest 2 mg daily for at least 6 months per os in combination with vaginal and rectal suppositories Longidaze® 1 suppository 1 time every 2 days 10 suppositories, and then 1 suppository 1 time in 7 days 17 suppositories for another 120 days;
5. Willingness to use barrier methods of contraception.

Exclusion Criteria:

1. Women before menarche or after menopause
2. Adenomyosis;
3. Amenorrhea (more than 3 months in a row within 6 months before screening);
4. Patients who are scheduled to undergo surgery for endometriosis during the study;
5. Hormone therapy for endometriosis or the use of aromatase inhibitors within 16 weeks prior to Day 0;
6. Daily use of pain relievers for 7 consecutive days or more due to any other reason other than endometriosis;

6. Participation in clinical trials less than 30 days before the screening visit and / or 5 drug half-lives, whichever is longer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a verified diagnosis of external genital endometriosis, who, as part of routine clinical practice, were prescribed monotherapy with per os dienogest or combined treatment with a combination of dienogest + vaginal and rectal suppositories Longidaze®, 3000 ME (hereinafter referred to as Longidaze® )
Sampling Method: Non-Probability Sample
Enrollment: 149 (Estimated)
Dates: Start 2019-12-26 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the severity of endometriosis-associated pelvic pain (Day 30) | Day 0, Day 30
  Changes in the severity of endometriosis-associated pelvic pain by visual analogue scale (VAS) after 30 days from the baseline value in patients of the dienogest + Longidaze® combination therapy group compared with patients who received only dienogest. The Visual Analogue Scale (VAS) is designed to measure pain intensity. It is a continuous scale in the form of a horizontal line 10 cm (100 mm) long and located on it two extreme points: "no pain" and "the strongest pain you can imagine." The patient is asked to place a line perpendicularly crossing the visual analogue scale at the point that corresponds to his pain intensity. The ruler measures the distance (mm) between "no pain" and "the worst pain imaginable," providing a score range from 0 to 100. A higher score indicates more pain intensity.

SECONDARY OUTCOMES:
Changes in the severity of endometriosis-associated pelvic pain (Days 90, 150, 180) | Day 0, Day 90, Day 150, Day 180
  Changes in the severity of endometriosis-associated pelvic pain according to the VAS after 90, 150 and 180 days relative to the baseline value in patients of the dienogest + Longidaze® combination therapy group compared with patients who received only dienogest. The Visual Analogue Scale (VAS) is designed to measure pain intensity. It is a continuous scale in the form of a horizontal line 10 cm (100 mm) long and located on it two extreme points: "no pain" and "the strongest pain you can imagine." The patient is asked to place a line perpendicularly crossing the visual analogue scale at the point that corresponds to his pain intensity. The ruler measures the distance (mm) between "no pain" and "the worst pain imaginable," providing a score range from 0 to 100. A higher score indicates more pain intensity.
Change in the Biberoglu and Berman scale | Day 0, Day 30, Day 90, Day 150, Day 180
  Change in the Biberoglu and Berman scale after 30, 90, 150 and 180 days from the baseline value from the start of treatment in patients of the dienogest + Longidaze® combination therapy group compared with patients who received only dienogest. The Biberoglu and Berman scale consists of five 4-point scales for assessing the severity of dysmenorrhea, dyspareunia and chronic pelvic pain not associated with menstruation, as well as the assessment of pain and static hyperalgesia during gynecological examination. In each of the scales, 0 points - no symptom, 3 points - the most pronounced symptom. The result is assessed by the sum of points for each symptom. With a sum of points from 1 to 2, pelvic pain is considered mild, from 3 to 5 - moderate, from 6 to 10 - strong, from 11 to 15 - severe.
Change in the score on the SF-36 quality of life questionnaire | Day 0, Day 30, Day 90, Day 150, Day 180
  Change in the score on the SF-36 quality of life questionnaire after 30, 90, 150 and 180 days relative to the baseline value from the start of treatment in patients of the dienogest + Longidaze® combination therapy group compared with patients who received only dienogest.
Change in the severity of uterine bleeding | Day 0, Day 30, Day 90, Day 150, Day 180
  Change in the severity of uterine bleeding after 30, 90, 150 and 180 days from the start of treatment in patients of the dienogest + Longidaze® combination therapy group compared with patients who received only dienogest. Patients will assess the severity of uterine bleeding in the patient's diary using the Mansfield-Voda-Jorgensen scale. There are five scoring options ranging from light bleeding to heavy bleeding. The rating is determined by the frequency of changing sanitary napkins or tampons, the degree of absorption of these products with blood, and also depends on the absorption properties of these products.

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - State budgetary healthcare institution "Chelyabinsk Regional Clinical Skin and Venereal Diseases Dispensary", Chelyabinsk, Chelyabinsk Oblast
  - Federal State Budgetary Scientific Institution "Research Institute of Obstetrics, Gynecology and Reproductology named after D.O. Ott ", Saint Petersburg, Leningradskaya Oblast'
  - Private health care institution "Road clinical hospital at the station Nizhny Novgorod of the open joint stock company" Russian Railways ", Nizhny Novgorod, Nizhny Novgorod Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Voronezh State Medical University named after N.N. Burdenko "of the Ministry of Health of the Russian Federation, Voronezh, Voronezh Oblast
  - Federal State Autonomous Educational Institution of Higher Education "Peoples' Friendship University of Russia", Moscow
  - Federal State Autonomous Educational Institution of Higher Education First Moscow State Medical University named after I.M. Sechenov of the Ministry of Health of the Russian Federation, Moscow

IPD SHARING:
Plan to Share IPD: No